CLINICAL TRIAL: NCT07358130
Title: Efficacies of Bismuth-amoxicillin-vonoprazan Triple Therapy and Bismuth Quadruple Therapy in the First-line Anti-Helicobacter Pylori Treatment
Brief Title: Efficacies of Bismuth-amoxicillin-vonoprazan Triple Therapy and Bismuth Quadruple Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Collaborators: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, DENG-CHYANG WU, Professor and Physician, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20250254
Record Dates: First submitted 2025-12-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori eradication
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Rabeprazole; Tetracycline; Metronidazole

STUDY DESIGN:
Intervention Model Description: bismuth-amoxicillin-vonoprazan triple therapy
Masking Description: bismuth-based quadruple therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bismuth-amoxicillin-vonoprazan triple therapy (Active Comparator): vonoprazan 20mg twice a day +tripotassium dicitrate bismuthate 300mg four times a day +amoxicilline 750mg four times a day
  Interventions: Drug: rabeprazole, tripotassium dicitrate bismuthate, tetracycline, metronidazole
- bismuth-based quadruple therapy (Active Comparator): rabeprazole 20mg twice a day+ tripotassium dicitrate bismuthate 300mg four times a day+ tetracycline 500mg four times a day+ metronidazole 250mg four times a day
  Interventions: Drug: vonoprazan, tripotassium dicitrate bismuthate, amoxicilline

INTERVENTIONS:
Drug: vonoprazan, tripotassium dicitrate bismuthate, amoxicilline — bismuth-amoxicillin-vonoprazan triple therapy
  Other Names: triple therapy
  Arms: bismuth-based quadruple therapy
Drug: rabeprazole, tripotassium dicitrate bismuthate, tetracycline, metronidazole — bismuth-based quadruple therapy
  Other Names: quadruple therapy
  Arms: bismuth-amoxicillin-vonoprazan triple therapy

SUMMARY:
(1) To compare the efficacy and safety of a 14-day bismuth-amoxicillin-vonoprazan triple therapy versus a 14-day bismuth-based quadruple therapy as first-line treatments for H. pylori infection, and (2) To investigate the influence of H. pylori antibiotic resistance, along with host CYP3A4, CYP2C19, and IL-1B -511 genotypes, on the eradication efficacy of H. pylori therapies.

DETAILED DESCRIPTION:
This multicenter, randomized, open-label, trial will enroll 552 adult patients with H. pylori infection from 12 medical centers or regional hospitals in Taiwan. Using a computer-generated randomization sequence (1:1 allocation; block size of four), participants will be assigned to receive either the 14-day bismuth-amoxicillin-vonoprazan triple therapy or the 14-day bismuth-rabeprazole-tetracycline-metronidazole quadruple therapy. Follow-up at week 2 will assess treatment adherence and adverse events. H. pylori status will be evaluated at week 6 using the C13-urea breath test. Eradication and adverse event rates will be compared between groups using the chi-square test. The impact of H. pylori antibiotic resistance and host CYP3A4, CYP2C19, and IL-1B -511 genotypes on treatment efficacy will be analyzed using multivariate models.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Helicobacter pylori infection

Exclusion Criteria:

1. Subjects with known hypersensitivity to the study drug.
2. Subjects with a history of gastric surgery.
3. Subjects with severe liver cirrhosis or uremia.
4. Subjects with a history of malignancy within the past five years.
5. Pregnant or breastfeeding women.
6. Subjects currently receiving treatment with atazanavir sulfate or rilpivirine hydrochloride.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of Helicobacter pylori eradication | 6 weeks after finishing study drugs
  evaluate eradication by 13C urea breath test
Evaluation of the safety of Helicobacter pylori eradication therapy | 14 days
  Drug-related adverse effects assessed by a standardized questionnaire

SECONDARY OUTCOMES:
genotype analysis | baseline
  Genotype analysis (CYP3A4, CYP2C19, and IL-1B -511) will be performed using a blood sample collected once at study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Deng-Chyang Wu, MD, PHD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No